CLINICAL TRIAL: NCT01597479
Title: Effectiveness of Distal Peripheral Nerve Blocks on Postoperative Pain Management After Ambulatory Thumb Resection Arthroplasty.
Brief Title: Ultrasound Guided Distal Peripheral Nerve Blocks and Postoperative Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-LEV-2011-21
Record Dates: First submitted 2012-05-07; First posted 2012-05-14 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Pain
Keywords: Ultrasound guided distal peripheral nerve blocks
MeSH Terms: conditions — Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No dPNBs group (No Intervention): Patients in this group didn't receive any intervention in the postoperative period.
- dPNBs group (Experimental): Patients in this group received ultrasound guided dPNBs on radial and median nerves (target nerves of TRA) in the postoperative period, before discharge.
  The procedural objective of dPNBs was to place local anesthetic around the target nerves to achieve a long lasting, sensitive and selective block in the surgical area. dPNBs were performed with 5 ml/nerve of levobupivacaine 0,125%.
  Ultrasound guidance allowed us to verify the correct distribution of LA around the target nerves target and optimize needle position if it was necessary, always avoiding the intraneural injection.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — In dPNBs group, we performed ultrasound guided dPNBs on radial and median nerves using low concentration and low volume of long acting local anesthetic (0.125% levobupivacaine, 5 ml per nerve). Using low concentrations of levobupivacaine on target nerves could achieve a prolonged sensitive block in the surgical area without motor block of the hand.
  Other Names: long acting local anesthetics
  Arms: dPNBs group

SUMMARY:
The aim of this clinical trial is to determinate if distal ultrasound guided peripheral nerve blocks on target nerves (radial and median nerve blocks at the elbow), using low volume and low concentration of long acting local anesthetic provide better postoperative pain control compare with systemic analgesia alone after thumb resection arthroplasty (TRA) due to a prolonged selective sensitive block on the tissue trauma.

DETAILED DESCRIPTION:
We designed a prospective randomized controlled trial, with nursing blinded evaluation.

We enrolled 52 patients scheduled for elective ambulatory TRA. 2 patients were excluded after randomization. Patients were randomized into two groups:

A. Group A= no distal peripheral nerve blocks (no dPNBs group; n = 24 ): We performed usual anesthetic technique for surgery: an AXILLARY BRAQUIAL PLEXUS BLOCK using SHORT ACTING local anesthetic (mepivacaine 1%). Patients allocated in this group didn't received any additional intervention in the postoperative period.

B. Group B (dPNBs group; n = 26): We performed the same anesthetic technique for surgery (AXILLARY BLOCK with 1% of mepivacaine) with an additional intervention. Patients allocated in this group received postoperatively dPNBs on target nerves. Based on surgical approached and technique we evaluated that radial and median nerves were responsible for the innervation of the surgical area, and therefore responsible for the postoperative pain. We performed dPNBs ON RADIAL AND MEDIAN NERVES (TARGET NERVES) WITH LONG ACTING AND LOW CONCENTRATION LOCAL ANESTHETIC (0,125% levobupivacaine 5ml/nerve).

All blocks were performed under ultrasound guidance.

Analgesic regime prescribed at discharge was the same in both groups: dexketoprofen with tramadol for rescue analgesia.

The primary outcome was to evaluate the proportion of patients experienced moderate to severe pain during first and second day postoperatively, mesured using a numerical visual scale (NVS) of 0 to 10 (0= no pain and 10= worst pain imaginable). We defined mild pain (NVS 0-3), moderate pain (NVS 7-10) and severe pain (NVS 7-10).

We considered dPNBs effective when patients experienced mild pain (NVS 0-3) for at least 6 hours after dPNBs puncture.

Secondary outcomes included:

1. Maximum pain intensity during first and second day postoperatively.
2. Duration of dPNBs, defined as the interval between dPNBs performance and the occurrence of first pain.
3. Time to discharge, defined as the interval since patient arrived at postoperative care unit (PACU) until discharge home.
4. Presence of distal hand motor block after dPNBs puncture.
5. Needed for rescue analgesia and total consumption of tramadol during first and second day postoperatively
6. Incidence of postoperative nausea and vomiting during 1st and 2nd day postoperatively
7. Needed for rescue antiemetic therapy, total consumption of ondansetron and effectiveness of treatment during 1st and 2nd day postoperatively.

Patients were contacted by phone first and second day postoperatively from a blinded PACU nursing staff (all outcome data were collected by PACU nursing staff blinded to group allocation).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years.
* Ambulatory TRA.
* Free acceptance to participate in the study, with informed consent signed by patient, guardian or family member.

Exclusion Criteria:

* Age less than 18 years
* Pregnancy.
* Inability to provide informed consent.
* Allergy to amide local anesthetics/NSAIDs
* Preexisting chronic pain treated with opioids.
* Neuropathy involving the extremity undergoing surgery or neurological-cognitive deficits that may interfere in the assessement.
* Contraindications to dPNBs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Rodriguez, anesthesia, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dufeu N, Marchand-Maillet F, Atchabahian A, Robert N, Ait Yahia Y, Milan D, Robert C, Coroir M, Beaussier M. Efficacy and safety of ultrasound-guided distal blocks for analgesia without motor blockade after ambulatory hand surgery. J Hand Surg Am. 2014 Apr;39(4):737-43. doi: 10.1016/j.jhsa.2014.01.011. Epub 2014 Feb 28. PMID 24582844
- [Background] Fredrickson MJ, Ting FS, Chinchanwala S, Boland MR. Concomitant infraclavicular plus distal median, radial, and ulnar nerve blockade accelerates upper extremity anaesthesia and improves block consistency compared with infraclavicular block alone. Br J Anaesth. 2011 Aug;107(2):236-42. doi: 10.1093/bja/aer101. Epub 2011 May 15. PMID 21576095
- [Background] Fredrickson MJ, Wolstencroft PJ, Chinchanwala S, Boland MR. Does motor block related to long-acting brachial plexus block cause patient dissatisfaction after minor wrist and hand surgery? A randomized observer-blinded trial. Br J Anaesth. 2012 Nov;109(5):809-15. doi: 10.1093/bja/aes266. Epub 2012 Aug 2. PMID 22864520
- [Background] Bouaziz H, Narchi P, Mercier FJ, Khoury A, Poirier T, Benhamou D. The use of a selective axillary nerve block for outpatient hand surgery. Anesth Analg. 1998 Apr;86(4):746-8. doi: 10.1097/00000539-199804000-00013. PMID 9539595
- [Background] Vial F, Bouaziz H, Mekler G, Cornet C, Merle M, Laxenaire MC. [Postoperative pain and surgical treatment of trapeziometacarpal osteoarthritis of the thumb after ambulatory surgery]. Ann Fr Anesth Reanim. 2000 Nov;19(9):643-8. doi: 10.1016/s0750-7658(00)00292-6. French. PMID 11244701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between february 2010 and april 2014, we enrolled 52 patients scheduled for elective ambulatory TRA under rutine axillary braquial plexus block.
Groups:
- Distal Peripheral Nerve Blocks Group (dPNBs Group): In dPNBs group, we practice distal peripheral nerves blocks guided by ultrasound and neurostimulator.
  Levobupivacaine: In dPNBs group, we practice ultrasound guided distal peripheral nerve blocks on radial and median nerves using low volume and low concentration of long acting local anesthetic (0.125% levobupivacaine, 5 ml per nerve).
  We performed dPNBs in the postoperative period. Deffered dPNBs under the influence of axillary block didn't cause patient disconfort. We considered the technique safety due to ultrasound guidance.
- No Intervention (no dPNBs Group): In patients of no dPNBs group didn't performed any intervention after surgery.
Period: Overall Study
Arm/Group | Distal Peripheral Nerve Blocks Group (dPNBs Group) | No Intervention (no dPNBs Group)
Started | 26 | 26
Completed | 24 | 26
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients undergoing Ambulatory TRA
Groups:
- dPNBs Group: dPNBs on radial and median nerves at the elbow in postoperative period, before discharge
- Non dPNBs Group: Non intervention in postoperative period
- Total: Total of all reporting groups
Arm/Group | dPNBs Group | Non dPNBs Group | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years]
  years | 67.4 (6.5) | 64.2 (7.5) | 65.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  Spain | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Experienced Moderate to Severe Pain During First and Second Postoperative Day
Description: Pain scores assessed using pain numerical visual scale (NVS) of 0-10 (o= no pain and 10= worst pain imaginable). We defined mild pain (NVS 0-3); moderate pain (NVS 4-6) and severe pain (NVS 7-10).The analysis of this variable at the end of the study will confirm or not the effectiveness of dPNBs for management of postoperative pain after TRA.
Time Frame: Up to 48 hours
Population: Patients undergoing ambulatory thumb resection arthroplasty (TRA)
Measure: Number; unit: percentage of patients
Groups:
- Distal Peripheral Nerve Blocks Group (dPNBs Group): We practiced ultrasound guided dPNBs on radial and median nerves, after surgery, before discharge.
  * Distal median nerve block was performed at the elbow, in the internal bicipital channel.
  * Distal radial nerve block was performed at approximately the junction of the middle and distal thirds of the arm.
  We use 5ml per nerve of levobupivacaine 0,125% for target nerve blocks.
- Non Distal Peripheral Nerve Blocks (Non dPNBs Group): Patients in non dPNBs didn't received any intervention in the postoperatively period.
Arm/Group | Distal Peripheral Nerve Blocks Group (dPNBs Group) | Non Distal Peripheral Nerve Blocks (Non dPNBs Group)
Number analyzed (Participants) | 24 | 26
percentage of patients
  Pain intensity NVS>3 on call 24h | 8.3 | 80.8
  Pain intensity NVS>3 on call 48h | 4.2 | 42.3

2. Secondary Outcome: Maximum Pain Intensity, Rescue Analgesia, Nausea and Vomiting Incidence, Use of Ondansetron for NVPO, Efectiveness of Ondansetron
Description: Number of participants with Maximum pain intensity NVS > 3; Rescue analgesia; Nausea and Vomiting incidence; use of ondansetron for NVPO; Ondansetron being effective (number of participants for whom ondansetron was effective to stop NVPO).
Time Frame: Up to 48 hours
Population: Patients undergoing ambulatory thumb resection arthroplasty
Measure: Number; unit: participants
Groups:
- dPNBs Group: we practiced ultrasound guided dPNBs on radial and median nerves using a long acting and low concentration local anesthetic (0.125% levobupivacaine, 5 ml per nerve).
- Non dPNBs Group: In this group any intervention was done.
Arm/Group | dPNBs Group | Non dPNBs Group
Number analyzed (Participants) | 24 | 26
participants
  Maximum pain intensity 24h (NVS>3) | 8 | 24
  Maximum pain intensity 48h (NVS >3) | 5 | 21
  Rescue analgesia 24h (n) | 2 | 17
  Rescue Analgesia 48h (n) | 5 | 17
  Nausea and vomiting 24h (n) | 1 | 10
  Nausea and vomiting 48h (n) | 0 | 5
  Use of ondansetron 24h (n) | 1 | 5
  Use of ondansetron 48h (n) | 0 | 5
  Effectiveness of ondansetron 24h | 1 | 4
  Efectiveness of ondansetron 48h | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Groups:
- Distal Peripheral Nerve Block Group: Any patient undergoing ultrasound guided distal peripheral nerve block reported any complication.
Arm/Group | Distal Peripheral Nerve Block Group
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

LIMITATIONS AND CAVEATS:
We could included another group: distal blocks with 0,125% levobupivacaine+ 4mg dexamethasone; register patient satisfaction with anesthetic technique or patient risks factors for nausea and vomiting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No